CLINICAL TRIAL: NCT06602102
Title: Pilot Study on Enhancing Mobility and Accessibility for Visually Impaired Individuals in Barcelona Using Navigation With XR Technology and 5G
Brief Title: Pilot Study on Improving Mobility and Universal Accessibility for Individuals With Visual Disabilities in Barcelona
Acronym: BCNMob
Status: Completed | Type: Observational
Sponsor: Universitat Politècnica de Catalunya (Other)
Responsible Party: Principal Investigator, Luis Perez, Clinical Professor, Universitat Politècnica de Catalunya
Other Study IDs: BCNMob; 22S07345-001 (Other Grant/Funding Number: La Caixa Foundation)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Low Vision Aids; Low Vision; Low Vision Blindness; Low Vision Digital Assistance
Keywords: low vision aids; low vision digital assistance
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low Vision: Participants with Low Vision
  Interventions: Device: Mixed reality Glasses

INTERVENTIONS:
Device: Mixed reality Glasses — Mixed reality glasses are devices that combine elements of augmented reality and virtual reality. They allow users to overlay digital images onto the real world, enabling interaction with virtual objects in a physical environment. These glasses typically use sensors, cameras, and tracking technology to map the surroundings and provide an immersive experience. They are used in various applications, such as gaming, education, design, and professional training.

SUMMARY:
The project BCNMob informs about a research study approved by the Ethics Committee of the Hospital Universitario Mútua Terrassa

The study aims to improve the Biel Glasses virtual reality glasses to assist patients with low vision in detecting and locating objects during mobility. Optometric evaluations and training sessions will be conducted, followed by tests in an urban environment in Barcelona.

There are no significant risks associated with participation, although mild discomfort may arise. The information collected will be confidential and managed according to data protection legislation. No financial compensation will be offered.

DETAILED DESCRIPTION:
Barcelona's Universal Accessibility Plan 2018-2026 is a commitment by the city to universal accessibility, regardless of people's condition.

Currently, the mobility problems of visually impaired people are mainly addressed through improvements in the accessibility of the space urban, the infrastructures, the facilities of use public i until i everything public transport.

Is calculated that the missing of autonomy staff generates one cost of more of €15,000/year for the people visually impaired. Also, studies show that 40% of visually impaired people fall once a year and 63% of these falls have medical consequences. The fear of suffering more falls causes social isolation, a sedentary behaviour and, consequently, a worsening of the quality of life, of the psychological state and of health in general, especially in the elderly, 10% of which can develop severe depression.

BCNMob project wants to contribute to reverse this situation, a thorough analysis and the measure of improving the mobility and universal accessibility of people with visual impairments in the city of Barcelona, through the development of devices with 5G technology in combination with artificial vision and augmented reality, integrated with the systems of Barcelona City Council&amp;amp;#39;s Open Data to inform users in real time.

The solution proposed by BCNMob is conceived from a perspective of collective and integrated use in the city, through a device sharing system that allows providing a mobility service adapted to the disability visual a so many people come be it possible, following one philosophy similar at service of "Bicing".

B. OBJECTIVES OF PROJECT AND QUESTIONS INVESTIGATION

The aim of the BCNMob project is to carry out a pilot study to analyse and measure the improvement of mobility and universal accessibility of people with visual impairments that can be achieved in the city of Barcelona, through the use of technology 5G in combination with other technologies such as artificial vision and augmented reality.

Nowadays, the mobility problems of visually impaired people are mainly addressed through improvements in the accessibility of the space urban, the infrastructures, the facilities of use public i until i everything public transport. Despite the undeniable usefulness of these measures, these actions do not allow by themselves the full mobility of these people, that they follow requiring of accompaniment for the carrying out the majority of their journeys, and who suffer from a strong dependence as a result of the lack of autonomy staff (see more forward, the section of Impact Social). How much the relationship of this problem with the objectives of the call, it must be taken into account that, due to the progressive nature of most of its causes, visual impairment affects the vast majority in the elderly, so according to WHO data, 80% of people who suffer from visual impairment are over 50 years old.

The project BCNMob pretends to change the shape to address this one problematic, posing more accent in the improving the ability of visually impaired people to move around like other people, allowing them to overcome by themselves the possible barriers that could limit their mobility and access to public spaces and services. However, the solution is conceived from a perspective of collective and integrated use in the city, through a system of sharing devices that allows providing a mobility service adapted to the visual impairment to as many people as possible, following a similar philosophy at service of Bicing . This one study will allow the validation of this technology come a possible solution that give answer to the requirements deployed by new Code of Accessibility of Catalonia, expected for this year 2022, and is aligned with the Barcelona Strategy for Universal Accessibility, which identifies the need to emphasize improvements in communicative accessibility (visual, sensory and cognitive).

To carry out the BCNMob project, the investigators will use technology developed by BIEL GLASSES SL (see details in the technology section). This technology has already been analysed and validated by the UPC in laboratory; Movilab; of the faculty of Optics i optometry of terrace (see removed of methodology, later). The Mobile World Capital foundation has selected Biel Glasses to carry out a first test of this technology during the month of July of this year the cities of Reus i Tarragona, come a case benchmark of how 5G technology can help people with disabilities, and has been awarded by the Agency Spatial European come one of the projects with greater potential that ago us of the European space technology.

The goals of the BCNMob project are much more ambitious, both from a technological point of view and from the analysis of the impact on the city and its inhabitants. So the investigators intend to move forward during the project in development of the state current of the technology for such to improve it the functionality, adding capacity of navigation adapted to people with visual impairments. The investigators also want to advance integration with the city itself, both technologically and socially: technologically through access to Open Data information relevant for the mobility of the people with disability visual, i with the training of system of AI to recognize the signage used in Barcelona; at a social level, through the realization of a first experience on an international scale of a device sharing system for improving autonomy of these people, front page a term in collaboration with the fabric associative represented for the Foundation period of view, entity integral of the table of accessibility of the network for the life Independent (XAVI) from Barcelona. Finally, the UPC&amp;amp;#39;s leadership will allow a scientifically accurate study to be carried out of the improvement achieved in mobility within the city and the accessibility of public spaces.

The specific objectives of the project are listed below, which will allow the achievement of the general objective of verifying whether the proposed technology can help the City of Barcelona improve the accessibility and mobility of people with visual impairments:

objectives of type technological

1. Develop the new functionalities of navigation adapted to the disability visual, combining i.a with the Galileo positioning system. Evaluation of the accuracy obtained in various areas of Barcelona with various architectural characteristics (existence of buildings that can block the satellite signal, narrow streets, etc.).
2. Integrate the information provided by the Open Data BCN service on works that may have an impact on the mobility of the people visually impaired, integrating it into the navigation system adapted
3. Fit the system to the characteristics specific to the city of Barcelona, including the necessary training of the system&amp;amp;amp;#39;s neural networks to guarantee the recognition of street crossing signage.
4. Assess the usability and reliability of the proposed technology, including aspects related to 5G coverage and the availability of EDGE, infrastructure within the city of Barcelona that allows the deployment of a technology like the one proposed.

Objectives related with the improvement of the mobility i the quality of life

1. to measure the improvement of the mobility i autonomy reached by participants in the study, a through of the KPI&amp;amp;#39;s that are defined for this purpose (see Methodology section).
2. evaluate the improvement in the accessibility of determined equipment/spaces public that will be included in the study, in agreement with Barcelona City Council.
3. evaluate the operation i the operability of the platform of use shared of the devices In this one section will be analysed come impact this one service of use shared the chain of accessibility of the spaces that will be included in the study, in accordance with the definition of this concept established in the Barcelona Strategy for Universal Accessibility 2022-2030. The accessibility chain of the proposed service will also be tested and analysed.
4. to spread the results of project BCNMob between the community scientific i divulge them between the collective of people with disability visual, like that come a level of the society in general i the administrations public
5. Contribute to better municipal decision-making in matters such as town planning, public space management, urban furniture, etc., following the results obtained in the mobility tests.

The questions the that Vol to give answer this one study are:

1. They allow new technologies such as 5G networks, Artificial Intelligence and Extended Reality to address the problem of mobility and universal accessibility of visually impaired people from a new perspective, improving their capabilities in order to equalize them with those of other people, allowing them to overcome by themselves the possible barriers that may limit their mobility and access to public spaces and services?
2. It is possible to design a device that, using these technologies, provides a level of usability, reliability, safety and comfort enough for such that the people with disability visual it adopts come a means to solve participants mobility problems and increase participants autonomy?
3. Is it possible to implement a service that makes this technology available to multiple users, sharing the necessary devices in a practical, effective, efficient and economically viable way? Within the framework of the project, the appropriate indicators (KPIs) will be designed to carry out the necessary measures to answer each of these questions objectively and well-founded.

   C. METHODOLOGY FORECAST

   According to the planned work plan, described in the schedule section, various methodologies will be used to carry out the various technical and scientific aspects of the project in each of its phases:

   PHASE 1. design and planning of the study pilot

   In this phase, the project&amp;amp;#39;s scientific team will determine the number and specific characteristics of users who can benefit from using the solution. The methodology to be used for the design and realization of the study is based on the conclusions obtained in the doctoral thesis of the Principal Investigator of the project."Design and implementation of a laboratory dedicated to the clinical validation of assistive technologies for perception and mobility in patients with peripheral field limitations", which refers to the laboratory; Movilab, built the facilities of the faculty of Optics i optometry of the UPC a Terrace, and what is one of the few two existing in Europe, which allows performing tests of technologies for the improvement of the mobility of visually impaired people, through the simulation of routes and situations where there are obstacles and other mobility risks. In this phase of the project this methodology will be adapted to the characteristics specific to project BCNMob, that is characterizing because the tests they will be carried out in locations in the urban environment of the city of Barcelona. Based on this methodology, the investigators will draw up a protocol that establishes the number of users, inclusion and exclusion criteria, optometric tests to be performed to assess their suitability, tests with the device and the metrics to be analysed. They are also included the statistical methods for the analysis of the results and ethical and data protection aspects and the times in which the project will be carried out are determined. This document will be presented to the Ethics Committee for approval before starting the tests. The most relevant aspects of this protocol are detailed below:
   * Design of the tests The design of the tests foresees one first phase for do essays in spaces exteriors, sure for the users, which will include sufficient elements relevant to mobility (obstacles, crossings, etc.). Afterwards, the assessment will be made in spaces/routes selected by the user, with the aim of assessing the level of impact of the mobility solution on their day-to-day life. In this phase, safety will be provided by accompanying a sighted guide. A coordination system will be designed between the escort and the user that allows the escort to stop the user before any situation of risk, without that this change the headquarters movement free i self-employed, for such of to allow to evaluate the improvement obtained.
   * determination of the variables of study i of headquarters register Systems will be implemented to control the parameters to be measured, both subjective (through the creation of surveys adapted to the study) and objective. For the various types of tests, quality markers (KPIs) will be defined, such as walking speed, recognition of the existence of obstacles, increase in distances travelled autonomously, decrease of hours of accompaniment, i also the measure of accessibility to certain equipment, system usability, etc. This information will be collected through user surveys.

   PHASE 2. recruitment of the candidates i the candidates

   - Diffusion of the study and contact with the possible candidates For the dissemination of the study, the investigators will use online and offline actions. Regarding online actions, the study will be published in the respective pages web of the entities that they form the consortium Also will be used the social networks. The Punt de Vista Foundation is very active on social networks (2000+ followers and speaker on various community platforms) and will coordinate the online dissemination of the BCNMob project, in its various stages how much the shares offline, the UPC will put in communication of the people candidates, between the users of the unity of come down vision of Centre university of the vision, where they receive attention patients that

   they gather the requirements for participate in the project on the other band, the Foundation period of view will spread the call between the professional community (College of Optics i optometrists (patron), Spanish Society of Baja Specialists Visión, etc.), health sector (IMO, Sant Joan de Déu, Sant Pau (Dr Díaz, patron), etc.), social sector and affected organizations (Associació Discapacitat Visual Catalunya B1B2B3 (patron), Retina Catalunya, ACIC, etc.) and networks public (Xavi, advice sectoral of people with disability, etc.). All these actions will be carried out respecting data protection legislation, avoiding unauthorized and indiscriminate communications at all times.

   - Characterization of the parameters visuals i functional of the participants with the goal of to determine the profile visual, theirs needs of mobility i the implications of acceptance of the solution technological, to the participants the study know them will perform one assessment visual functional (binocular) of visual acuity, visual field, contrast sensitivity, glare recovery time and color vision, as well as the collection of information on the present time of the disability and the reflex in the resolution of activities of daily living

   PHASE 3. development i integration
   * technology object of the study The technology that aims to evaluate the project BCNMob is developed for BIEL GLASSES SL This company is the result of the initiative of the parents of Biel, a child with congenital visual impairment who suffers from mobility limitations as a result of his disability. His parents, a doctor and an electronic engineer, decided to start the project when they saw that there were no solutions on the market that would allow Biel to move around the city autonomously and safely.

   The system is based on a device consisting of smart glasses that solve the users&amp;amp;amp;#39; mobility problems using a combination of the most advanced technologies (AI - Artificial Intelligence, robotics, XR- reality extended, 5G i geolocation Galileo). These glasses are able to understand reality and adapt it to the user&amp;amp;amp;#39;s ability to perceive for such that can move around of shape autonomous The device detects mobility risks such as obstacles, steps, holes, pedestrian crossings or traffic lights, and uses XR for insert in the image directions graphics adapted to the remaining vision of each patient. In addition, the system incorporates a navigation system of high accuracy based on in the combination of AI i the system of Galileo positioning, which provides directions adapted in the same way. In the following video, one can see an explanation of how the device works:https://vimeo.com/465500260

   The device uses 5G technology to connect to the platform at cloud for such of power bring a term the high computational load processes that are required. The large bandwidth of 5G and its low latency make it possible to do these tasks in the cloud without reduce the quality of the image and reaction times, which is absolutely critical in an application come this one The consequent reduction of the load of the local processor of the device allows reducing its consumption of energy, the weight, the size i the cost For reduce even more latency, technology is used, which brings the infrastructures closer together of computation the border of the network 5G. The fault-tolerant design maintains the ability to locally perform safety-critical functions, such as obstacle detection, in the event of a 5G connection loss.

   The 5G connection allows also the access resources in line come bases of cartographic data necessary for the navigation In this one meaning, come a party of project it foresees to include the integration of system with the platform ;Open date BCN; for such to access an information updated about works have to place the city of Barcelona that they can make it difficult the displacement of the users The system will use this one information both to warn users when they are approaching, and to calculate routes so that they can be avoided. Thank you at headquarters design based on in XR, the system no only is capable of to provide directions adapted to the user&amp;amps visual capacity, but also allows working on the image itself to offer visual improvements such as zoom vision or dynamic light adaptations, to avoid glare and night blindness, very common in people with problems of peripheral visual field.

   The solution includes a platform also based on the cloud that allows that the devices be used by multiple users by automatically downloading the configuration of each of them. The configuration for each patient is performed only once by one optometrist, this allows to get the maximum performance of the vision that the user retains. From then on, the system stores this configuration to be downloaded to any device that the user person needs to use. The system provides for the use of cabins of collection and deliver sanitized, for the which thing the model of use shared of devices may be implemented in urban areas by public health systems, social services or associations/foundations related with the disability visual The delivery of the device's address can also be implemented according to the preferences and capabilities of the institutions providing the service, including the sanitation process.

   - Tests : Before using the device with users, the investigators will perform validation tests of the device's technical functions in the MoviLab laboratory environment.

   - Methodology of management of project technological This phase includes the development and integration tasks that must allow the use of the technology developed by BIEL GLASSES for the realization of the BCNMob project. These tasks make up one project technological inside of project general of pilot, i in consequence, for bring it a term the investigators will use project management methodology, to achieve the planned objectives within the pre-established term i with budgeted costs. The management team of project will maintain communication between all interested parties in the project and identify deviations in the Project Plan with respect to its development in the three slopes of the management of projects: scope of realization or reach of goals, execution term and costs incurred during everything the project is will last a term one tracking of same with the aim of coordinating the work of the different teams involved, compiling all the results obtained, determining the decisions to be made at each stage of the project and establishing the appropriate priorities.

   Likewise, will take care of maintenance of the documentation generated in the project, including the reports and correspondence. He will also draw up the meeting minutes of the Project Management Committee and keep the rest of the researchers informed, both from his own group and of the collaborators. The meetings of the Project Management Committee will be convened periodically in order to monitor and verify the fulfilment of its objectives, to correct any deviations that may have arisen and to plan the work to be carried out according to the planning established temporary Risk management will also be one of the fundamental parts of the Project Management Committee. During execution of project, for a minimize anyone risk additional no expected, they will identify themselves some of the more risks important of project i the headquarters possible plan of contingency The responsible for project will be the person in charge of the evaluation continuous of the management of risk, like that come of the update of the analysis of risks and of plan of contingencies depending on the results that are consumed during the project. The risk management plan for the project is shown in the adjacent figure.

   In relation to the software development that is necessary for the adaptation of the technology to the objectives of the pilot study, SCRUM methodologies will mainly be used.

   PHASE 4. execution of pilot
   * Shares formative

   The investigators will three type of shares trainings:

   - Training of the people companions (guides seers), for to allow the coordination with the user person during the tours, for to manage the risks without alter the headquarters movement free i autonomous and facilitate the evaluation of the improvement obtained;
   * Training in the usability of the devices for people users i technicians;
   * Operation of the platform of use shared to the people users, companions and technicians
   * Tests of mobility i universal accessibility How it has indicated previously, for the execution of this phase will be used the methodology developed by the Principal Investigator in her doctoral thesis, modified during the design phase in order to adapt it to the requirements of the proposed study. A noteworthy aspect of this methodology is the use of observers simulators The observers simulators they are people with vision normal that they use simulation systems to restrict their vision similarly to that of the visually impaired. The participation of these people will allow doing one validation of the areas of tests before of the participation of the members of the study cohort. This validation includes both the aspects related to the relevance and adequacy of the tests with respect to the indicators a measure, come the safety of the members of the cohort The results obtained will serve to make adjustments or improvements in the design of the study.

   PHASE 5. analysis of the tests carried out

   - Analysis i conclusions of the results obtained They will be analysed so much the results measurable of shape objective (reduction of collisions, reduction of the time required to complete the routes, etc.) as well as the subjective opinions of the users (satisfaction, usability of the system, etc.).

   - Proposal of improvements in the system

   PHASE 6. Shares of disclosure to see removed specific of Actions of disclosure (section J). Projects network communication, as well as the creation of associated audiovisual resources, will be carried out by Silvia Martín, communication technician at the Punt de Vista Foundation.

   D. RESULTS The investigators hope that the results of the study will allow us to confirm an increase in the autonomy of visually impaired people who use the system, of at least 85%, measured as the increase in routes that is they can perform of shape autonomous this one indicator will form party of one set a lot more complete that must allow measuring and, where appropriate, validate the usefulness of technology both to improve mobility and the accessibility of urban spaces. The investigators also hope to extend the current functionalities of the system, including the capacity of navigation adapted i the integration with the information &amp;amp;amp;#34;Open date&amp;amp;amp;#34; offered by Barcelona City Council, to be able to provide full autonomy to users. Finally, the investigators hope to validate the usability, reliability and security of the technology, to the point where the investigators can ensure the success of a potential deployment.

   For that ago the citizenship, these results they have of to allow advance in the development i deployment of technologies that allow the improvement of mobility and the quality of life of people with visual impairments, especially of the people great that in suffer, that in they are the big majority of the affected These people add to the mobility and quality of life problems generated by visual impairment, their own physical and social fragility can lead to more severe consequences when accidents or disorientation occur, such as social isolation caused by the fear of suffering, which significantly impacts their quality of life (see the Social Impact section).

   For that ago the decisions policies, is clear that these they will be necessary for materializing the advances that can facilitate the technology, i too it will be that is they can to take of shape grounded the investigators wait that the results of the study provide sufficient evidence to consider this technology among the options a have in account for the improvement of the mobility and the quality of life of the people with visual impairment a Barcelona, with special attention the people great affected In specific, the investigators wait that the results are they can to have in account in the implementation of the Strategy Barcelona for Accessibility universal 2022-2030 and to comply with the next Accessibility Code of Catalonia.

   Regarding knowledge, it is important to bear in mind that this technology is fully developed in Barcelona, by a company that is also being incubated by Barcelona Activa, having been selected to participate in several programs of this entity as an of the projects with major potential so much at a technological level like social it is of course the results of this project will contribute in form decisive the improvement i validation of this technology and am the consolidation of the company, i that the results of this study they will serve of reference a level international for the possible extension an others cities of Europe and beyond, contributing at growth of Barcelona come a referent technological i too at growth of technological sector in areas of maximum interest for its innovation such as artificial intelligence, extended reality, applications of 5G networks and robotics.

   E. CHRONOGRAPH

   Below is the work plan in its various phases, associated tasks and responsibilities (UPC for Universitat Politècnica de Catalunya, BG for Biel Glasses SL and PDV for the Punt de Vista Foundation) and the schedule:

   I. JUSTIFICATION OF THE ADVANTAGES FROM LA COOPERATION OF THE APPLICANTS BCNMob project team is made up of experts in the fields of optometry, medicine, technology, scientific dissemination and management which, together, bring more than 50 years of experience in the field of Information Technologies and 30 years in medical research and visual health.

   The achievement of the objectives that is raises the project BCNMob is possible only thank you to the synergies generated between the three entities that make up the consortium. Their complementarity is based on the areas of contrasting expertise of each and on the history of previous collaborations between the three organizations, and constitutes the starting point of the BCNMob project, its main asset and the added value of the initiative.

   J. IMPACT SOCIAL FROM LA RESEARCH

   For a understanding the impact social i economic of project BCNMob about the people with come down vision (BV) it is necessary to understand the impact that mobility problems have on these people, and that can be divided into tangible and intangible aspects. Here are the tangibles:

   - The missing of autonomy carries problems of dependency

   - From the labour point of view, mobility problems mean that the offer of jobs to people with disabilities visual be in the immense majority places that no they involve mobility, the which thing reduces supply and has an impact on a very high unemployment rate (over 75% in 2019, according to data from the European Blind Union).

   - Lack of autonomy combined with deteriorating health (see intangible effects below) can behave in the institutionalization of the person, the which thing is a lot expensive and involves other risks, as demonstrated by the COVID-19 pandemic.

   Economically, existing estimates calculate the combined impact of tangible aspects at approx €15,000/year/person a Europe 1 (costs adjusted to the inflation), being the costs of dependence and institutionalization the highest.

   The aspects of intangibles, still that no less important, include the following:
   * The mobility reduced implies the incapacity to maintain and generate relationships outside of one environment local i the close family circle, causing social exclusion.

ELIGIBILITY:
Inclusion criteria:

* Minimum age of 18 years.
* Patients with peripheral vision (PV) <20º in both eyes, and the patient expresses difficulty in their ability to move independently and safely in everyday environments.
* Distant visual acuity with the best possible correction in the better eye (VA) ≤ 0.3 (30%) and who expresses problems orienting in external environments.

The use of a cane or any other mobility aid is NOT an exclusion criterion.

* Patients with ophthalmological diagnoses: glaucoma, retinitis pigmentosa, Leber congenital amaurosis, high myopia, diabetic retinopathy, and other pathologies that cause hemianopsias.
* Ability to understand and follow the study instructions.
* Physical and cognitive ability to use virtual reality glasses and actively participate in the tests.
* Availability to participate in the study (8 hours on average spread over 3-4 sessions).
* The tests to evaluate the patien';s visual examination will be conducted at the Centre Universitari de la Visió (CUV) CUV Terrassa: Passeig del Vint-i-dos de Juliol, 660, 08222 Terrassa.

Exclusion criteria:

* Patients who are in active treatment for ocular conditions or who have received recent ophthalmological treatment or have had prior surgery within 3 months before the start of the study tests.
* Patients diagnosed with neurodegenerative diseases.
* Presence of medical or psychological conditions that may interfere with the safe participation in the study.
* Individuals who have difficulties moving independently due to a condition or pathology unrelated to their visual ability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this research will consist of individuals who meet the inclusion and exclusion criteria, belonging to the metropolitan area of Barcelona.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Number of obstacles identified in time and avoided | Throughout the testing session with the virtual reality glasses.
  The number of obstacles present in the urban circuit that the participant detects and successfully avoids will be measured
Walking speed while using virtual reality (VR) glasses | From enrollment to the end of treatment at 2 weeks
  The walking speed of the participants will be measured while wearing virtual reality glasses in an urban environment.

SECONDARY OUTCOMES:
Number of obstacles touched | From enrollment to the end of treatment at 2 weeks
  The number of obstacles the participant has collided with while wearing the virtual reality glasses.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Gispets, PhD, Principal Investigator — Universidad Politécnica de Catalunya; Salut Alba-Arbalat, PhD, Study Chair — Universidad Politécnica de Catalunya
Locations (1):
- Facultad de Óptica y Optometría de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The data from this study cannot be shared with others for several reasons. Firstly, this is a pilot observational study aimed at collecting a specific set of data to improve the evaluated tool. The primary focus is on refining the methodology and understanding preliminary outcomes, rather than generating widely shareable results.
  Secondly, the data collected in this pilot phase is intended to inform a future, more comprehensive study. In that subsequent study, we plan to evaluate the effectiveness of the tool more rigorously, at which point data sharing may be considered appropriate.
  Finally, sharing data at this stage could compromise the integrity of the study and the validity of future research. Therefore, it is crucial to maintain the confidentiality and exclusivity of the data until the final study is conducted.

REFERENCES:
- [Background] Resnikoff S, Pascolini D, Etya'ale D, et al. Global data on visual impairment in the year 2002. Bull World Health Organ 2004; 82: 844-851. Peters D, Bengtsson B, Heijl A. Lifetime risk of blindness in open-angle glaucoma. Am J Ophthalmol 2013; 156: 724-730. Bourne RRA, Flaxman SR, Braithwaite T, et al. Magnitude, temporal trends, and projections of the global prevalence of blindness and distance and near vision impairment: a systematic review and meta-analysis. Lancet Glob Health 2017; 5: e888-e897. Bourne R, Price H, Taylor H, et al. New systematic review methodology for visual impairment and blindness for the 2010 Global Burden of Disease study. Ophthalmic Epidemiol 2013; 20: 33-39. Burton MJ, Ramke J, Marques AP, et al. The Lancet Global Health Commission on Global Eye Health: vision beyond 2020. Lancet Glob Health 2021; 9: e489-e551. Wang MY, Rousseau J, Boisjoly H, et al. Activity limitation due to a fear of falling in older adults with eye disease. Invest Ophthalmol Vis Sci 2012; 53: 7967-7972. Kempen GIJM, Ballemans J, Ranchor AV, et al. The impact of low vision on activities of daily living, symptoms of depression, feelings of anxiety and social support in community-living older adults seeking vision rehabilitation services. Qual Life Res 2012; 21: 1405-1411. Wang MY, Rousseau J, Boisjoly H, et al. Activity limitation due to a fear of falling in older adults with eye disease. Invest Ophthalmol Vis Sci 2012; 53: 7967-7972. Ong SR, Crowston JG, Loprinzi PD, et al. Physical activity, visual impairment, and eye disease. Eye 2018; 32: 1296-1303. Steinberg EP, Tielsch JM, Schein OD, et al. The VF-14. An index of functional impairment in patients with cataract. Arch Ophth